CLINICAL TRIAL: NCT01160861
Title: A Phase Ib, Randomized, Blinded, Placebo-Controlled, Multiple-Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of MEMP1972A in Patients With Allergic Rhinitis
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of MEMP1972A in Patients With Allergic Rhinitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MOP4840g
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- A (Experimental)
  Interventions: Drug: MEMP1972A; Drug: placebo
- B (Experimental)
  Interventions: Drug: MEMP1972A; Drug: placebo
- C (Experimental)
  Interventions: Drug: MEMP1972A; Drug: placebo

INTERVENTIONS:
Drug: MEMP1972A — Repeating ascending dose
Drug: placebo — Repeating ascending dose

SUMMARY:
This is a Phase Ib, randomized, blinded, placebo-controlled, multiple-ascending dose study in patients with seasonal or perennial allergic rhinitis to investigate the safety, tolerability, and pharmacokinetics (PK) of MEMP1972A.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of allergic rhinitis
* In good health, determined by no clinically significant findings from medical history, 12-lead ECG, and vital signs
* Males or females who are surgically sterilized, post menopausal for the past year, or are using two acceptable methods of contraception against pregnancy through at least 6 months after the dose of study drug

Exclusion Criteria:

* History or clinical manifestations of significant metabolic, hepatic, renal, hematologic, immunodeficiency, pulmonary, cardiovascular, gastrointestinal, urologic, neurologic, or psychiatric disorders
* History of anaphylaxis, hypersensitivity or drug allergies
* Use of a non-biologic investigational drug or participation in an investigational study with a non-biologic drug within 30 days prior to dosing
* Use of a biologic investigational therapy or participation in an investigational study involving biologic therapy within 3 months prior to dosing
* Positive blood test for chronic viral infections by: hepatitis B surface antigen, hepatitis C virus antibody, or HIV antibody

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-07-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of laboratory abnormalities, based on hematology, clinical chemistry, and urinalysis test results | Throughout study or until early discontinuation
Incidence, nature, and severity of adverse events | Throughout study or until early discontinuation

SECONDARY OUTCOMES:
Pharmacokinetic parameters of MEMP1972A (maximum plasma concentration, total serum clearance, volume of distribution, half-life) | Throughout study or until early discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Harris, M.D., Ph.D., Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Gauvreau GM, Harris JM, Boulet LP, Scheerens H, Fitzgerald JM, Putnam WS, Cockcroft DW, Davis BE, Leigh R, Zheng Y, Dahlen B, Wang Y, Maciuca R, Mayers I, Liao XC, Wu LC, Matthews JG, O'Byrne PM. Targeting membrane-expressed IgE B cell receptor with an antibody to the M1 prime epitope reduces IgE production. Sci Transl Med. 2014 Jul 2;6(243):243ra85. doi: 10.1126/scitranslmed.3008961. PMID 24990880